CLINICAL TRIAL: NCT01978665
Title: The Effect of Prednisone and Solu-Medrol on Physical Exercise in COPD Patients and the Inflammaroty Response During and After Exercis.
Brief Title: The Effect of Prednisone on Physical Exercise in COPD Patients
Acronym: COPDpred
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Bispebjerg Hospital (Other)
Responsible Party: Principal Investigator, Vibeke Backer, professor, Bispebjerg Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 2012-004503-13; 2012-004503-13 (EudraCT Number)
Record Dates: First submitted 2013-11-01; First posted 2013-11-07 (Estimated); Last update posted 2020-02-05 (Actual); Status verified 2013-11

CONDITIONS: Exercise Performance in Copd Patients
Keywords: COPD exercise inflammation prednisone
MeSH Terms: interventions — Prednisone

STUDY DESIGN:
Intervention Model Description: RCT study with steroid.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- prednisone and Solumedrol (Placebo Comparator): placebo arm versus prednisone
  Interventions: Drug: prednisone
- solumedrol (Placebo Comparator): placebo versus solu medrol
  Interventions: Drug: prednisone
- placebo (Other): measurement of fitness
  Interventions: Drug: prednisone

INTERVENTIONS:
Drug: prednisone — similar size tablets
  Other Names: placebo

SUMMARY:
The objective of this study is to investigate if there is an effect on exercise performance og of the anti inflammatory drugs prednisone and solu-medrol in patints with chronic obstructive pulmonary disease(COPD)

DETAILED DESCRIPTION:
RCT study with 4 days of steroid

ELIGIBILITY:
Inclusion Criteria:FEV1< 60% FEV1/FVC ratio <70 %

* able to use a ergometer bike

Exclusion Criteria: Haemodynamicaly unstable heart conditions

* exacerbations before 6 week entry of the study exacerbation during the study period treatment with beta blockers malignancy the last 5 years allergi toward IMP

Ages: 40 Years to 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2013-04 (Actual); Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
effect on muscle power | jan 2013 to july 2013 (6 months)
  muscular strenght

SECONDARY OUTCOMES:
the inflammatory response | jan 2013 to july 2013 (6 months)
  hsCRP

OTHER OUTCOMES:
vo2max | jan 2013 to july 2013 ( 6 months)
  fitness
VO2max | jan 2013 until july 2013 (6 months)
  fitness

CONTACTS AND LOCATIONS:
Overall Officials: Vibeke Backer, professor, Principal Investigator — Bispebjerg Hospital
Locations (1):
- Bispebjerg Hospital, Copenhagen, NV, Denmark